CLINICAL TRIAL: NCT00425594
Title: A Safety and Efficacy Evaluation of 3 Bowel Preparations in the Pediatric Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: John McGowan, Clinical Operations Manager, Braintree Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F38-25
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Colonoscopy
Keywords: colonoscopy; bowel preparation; prep
MeSH Terms: interventions — Bisacodyl; polyethylene glycol 3350

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: HalfLytely and Bisacodyl Tablets - Formulation 1
Drug: HalfLytely and Bisacodyl Tablets - Formulation 2
Drug: NuLYTELY

SUMMARY:
This randomized, parallel, multi-center, single-blind study is designed to compare the safety and efficacy of 3 bowel preparations in pediatric subjects scheduled to undergo a colonoscopy for a routinely accepted indication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are undergoing colonoscopy for a routinely accepted indication, including:

  * Evaluation of BE results
  * Endosonography
  * Blood in stool
  * Anemia of unknown etiology
  * Abdominal Pain
  * Polypectomy
  * Unknown diarrhea or constipation etiology
  * Inflammatory bowel disease
* Between 6 and 16 years of age at screening.
* Otherwise in good health, as determined by physical exam and medical history.
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, sterilized, abstinent, or vasectomized spouse).
* Negative urine pregnancy test at screening, if applicable
* In the investigator's judgment, parent/guardian is mentally competent to provide informed consent to participate in the study.

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, or toxic megacolon
* Subjects impacted at screening
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects who are undergoing colonoscopy for foreign body removal and decompression
* Subjects with known difficulties for swallowing tablets
* Subjects with pre-existing electrolyte disturbances, such as dehydration, or those secondary to the use of diuretics.
* Subjects who are taking drugs that may affect electrolyte levels with the exception of routine diuretics.
* Subjects with known clinically significant electrolyte abnormalities such as hypernatremia, hyperphosphatemia, hypokalemia, or hypocalcemia
* Subjects who are pregnant or lactating, or intending to become pregnant during the study.
* Subjects of childbearing potential who refuse a pregnancy test.
* Subjects who are allergic to any preparation components
* Subjects who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days.
* Any condition in parent/guardian associated with poor subject compliance (e.g., substance abuse); inability of parent/guardian to return for scheduled visits with their child.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Efficacy - preparation quality using a 4-point scale

SECONDARY OUTCOMES:
Safety - patient reported preparation related side effects. Pre and post preparation analysis of serum chemistry.

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (26):
- United States (26):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Tuscaloosa, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - San Francisco, California
  - Gainesville, Florida
  - Orlando, Florida
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Morristown, New Jersey
  - Buffalo, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Lancaster, Pennsylvania
  - Columbia, South Carolina
  - Houston, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Milwaukee, Wisconsin